CLINICAL TRIAL: NCT07235163
Title: AN INTERVENTIONAL, PHASE 1, RANDOMIZED STUDY WITH DOUBLE-BLIND AND SPONSOR-OPEN, PLACEBO-CONTROLLED SINGLE AND MULTIPLE DOSE ESCALATION TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND IMMUNOGENICITY OF PF-08065010 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-08065010 Are Tolerated and Act in the Body of Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C6341001
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part A: Cohort 1: single ascending dose (SAD) (Experimental): Dose A - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 2: single ascending dose (SAD) (Experimental): Dose B - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 3: single ascending dose (SAD) (Experimental): Dose C - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 4: single ascending dose (SAD) (Experimental): Dose D - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 5: single ascending dose (SAD) (Experimental): Dose E - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 6: single ascending dose (SAD) (Experimental): Dose F - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 7: single ascending dose (SAD) (Experimental): Dose G - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 8: single ascending dose (SAD) (Experimental): Optional Japanese Cohort dose to be determined - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 9: single ascending dose (SAD) (Experimental): Optional Chinese Cohort dose to be determined - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 10: single ascending dose (SAD) (Experimental): Optional Cohort with dose to be determined - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part A: Cohort 11: single ascending dose (SAD) (Experimental): Optional Cohort with dose to be determined - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part B: Cohort 12: multiple dose (Experimental): Dose F - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part B: Cohort 13: multiple dose (Experimental): Optional Cohort with dose to be determined - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo
- Part B: Cohort 14: multiple dose (Experimental): Optional Cohort with dose to be determined - Participants will receive PF-08065010 or placebo.
  Interventions: Drug: PF-08065010; Drug: Placebo

INTERVENTIONS:
Drug: PF-08065010 — Experimental Pfizer compound which will be subcutaneous (SC) or intravenous (IV).
Drug: Placebo — Placebo which will be SC or IV

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (called PF-08065010) for possible treatment of rheumatoid arthritis (RA) and systemic lupus erythematosus (SLE).

This study is seeking participants who are:

* male or female between 18 and 65 years of age
* deemed to be healthy

Participants in this study will receive PF-08065010 or placebo. A placebo does not have any medicine in it but looks just like the medicine being studied. PF-08065010 or placebo will be given as a shot (in the abdomen, thigh or back of the arms) or as an IV infusion in the arm (given directly into a vein) at the study clinic.

In Part A, participants will take PF-08065010 or placebo only 1 time and will take part in this study for about 5 months. During this time, they will stay at the study clinic for about 9-10 days and will have about 6 more study visits at the study clinic.

Participants in Part B of the study will take PF-08065010 or placebo once a month, for 3 months and will take part in this study for about 7 months. During this time, they will stay at the study clinic for about 4 days each month and will have about 6 more study visits at the study clinic.

During study clinic stays and study visits, urine, blood samples, and physical exams will be done.

ELIGIBILITY:
Inclusion Criteria:

* male or female between 18 and 65 years of age
* deemed to be healthy

Exclusion Criteria:

1. Evidence or history of clinically significant medical conditions.
2. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg)or hepatitis C antibody (HCVAb).
3. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
4. A positive urine drug test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-04 (Estimated); Primary Completion 2027-06-09 (Estimated); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline, approximately up to 5 months
  Part A
Number of Participants With Clinically Significant Laboratory Abnormalities | Baseline, approximately up to 5 months
  Part A
Number of Participants With Vital Sign Abnormalities | Baseline, approximately up to 5 months
  Part A
Number of Participants with Change from Baseline in Physical Exam (PE) Parameters | Baseline, approximately up to 5 months
  Part A
Number of Participants with Change from Baseline in Electrocardiogram (ECG) Parameters | Baseline, approximately up to 5 months
  Part A
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline, approximately up to 7 months
  Part B
Number of Participants With Clinically Significant Laboratory Abnormalities | Baseline, approximately up to 7 months
  Part B
Number of Participants with Vital Sign Abnormalities | Baseline, approximately up to 7 months
  Part B
Number of Participants with Change from Baseline in Physical Exam (PE) Parameters | Baseline, approximately up to 7 months
  Part B
Number of Participants with Change from Baseline in Electrocardiogram (ECG) Parameters | Baseline, approximately up to 7 months
  Part B

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Profile from Time Zero to the Time of Last Quantifiable Concentration (AUClast) | Predose (Day 1), approximately up to 5 months
  Part A
Area Under the Curve from Time Zero to Extrapolated Infinite Time (AUCinf) | Predose (Day 1), approximately up to 5 months
  Part A
Maximum Observed Plasma Concentration (Cmax) | Predose (Day 1), approximately up to 5 months
  Part A
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose (Day 1), approximately up to 5 months
  Part A
Plasma decay half-life (t1/2) is the time measured for the plasma concentration to decrease by one half. | Predose (Day 1), approximately up to 5 months
  Part A
Area under the serum concentration time profile over the dosing interval of 28 days (AUCtau) | Predose (Day 1), approximately up to 7 months
  Part B
Maximum Observed Plasma Concentration (Cmax) | Predose (Day 1), approximately up to 7 months
  Part B
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose (Day 1), approximately up to 7 months
  Part B
Plasma Decay Half-Life (t1/2) | Predose (Day 1), approximately up to 7 months
  Part B

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6341001